CLINICAL TRIAL: NCT05529056
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Therapeutic Effect and Safety of LPTAT in Children With Myopia
Brief Title: Study of Atropine Therapeutic Effect on Myopic Progression
Acronym: STAMP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: LitePharmTech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LPT-01
Record Dates: First submitted 2022-08-10; First posted 2022-09-06 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Myopia; Children
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Test Arm 1 (Experimental): LPTAT01
  Interventions: Drug: Atropine Sulfate 01
- Test Arm 2 (Experimental): LPTAT02
  Interventions: Drug: Atropine Sulfate 02
- Test Arm 3 (Experimental): LPTAT03
  Interventions: Drug: Atropine Sulfate 03
- Reference Arm (Placebo Comparator): LPTAT04
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atropine Sulfate 01 — Atropine sulfate 01 ophthalmic solution
  Other Names: LPTAT01
  Arms: Test Arm 1
Drug: Atropine Sulfate 02 — Atropine sulfate 02 ophthalmic solution
  Other Names: LPTAT02
  Arms: Test Arm 2
Drug: Atropine Sulfate 03 — Atropine sulfate 03 ophthalmic solution
  Other Names: LPTAT03
  Arms: Test Arm 3
Drug: Placebo — Placebo ophthalmic solution
  Other Names: LPTAT04
  Arms: Reference Arm

SUMMARY:
This study is to evaluate the therapeutic effect and safety of LPTAT in children with myopia.

DETAILED DESCRIPTION:
The primary objective is to evaluate the superiority of LPTAT to placebo in slowing myopia progression through the change of SE(Spherical Equivalent), which is measured by cycloplegic autorefraction after 12-month treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 5 to 12 years at the time of consent
* Refractive error of SE at least -1.0 D and no greater than -8.0 D in both eyes as measured by cycloplegic autorefraction at visit 1 and visit 2.
* Confirmed myopia progression of 0.5D or more within past 1year
* Astigmatism of 2.5D or less in both eyes
* Distance Best Corrective Visual Acuity to logMAR 0.2 or better in both eyes at visit1.
* Normal IOP under 21mmHg in both eyes.
* Anisometropia of SE less than 2.0D as measured by cycloplegic autorefraction at visit 1.
* Written informed consent willingly obtained by both subject and his/her parents

Exclusion Criteria:

* Hypersensitivity to atropine or other cycloplegic agent.
* History of the surgery of refractive correction
* Having ocular disease affect to visual function or refractive error: history of glaucoma, macula r degeneration, diabetic eye disease, uveitis, etc, or presence of conjunctivitis at screening visit.
* Having systemic diseases that affect to vision loss
* Having risk of IOP elevation such as narrow angle, Shallow Anterior Chambers, etc
* Presence of binocular function disorder or stereopsis disorder
* Amblyopia or manifest strabismus
* History of premature birth(less than 37weeks) or low birth weight(less than 2,500g)
* Previous or current use of atropine or Ortho-K lens for myopia
* Down syndrome, spastic paralysis, brain damage, spastic palsy, bladder
* Presence of neurological diseases like epilepsy, etc. which could expect difficulties in compliant to the ocular examinations.
* Presence of clinically significant cardiac and respiratory diseases
* Participation in any other clinical study of an investigational product within 3-month prior to current IP administration.
* Based on the investigator's discretion, subject who is not proper to participate in the trial.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 472 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Spherical Equivalent over 12-month | 12 months
  Change in spherical equivalent measured by cycloplegic autorefraction at 12 months after administration of clinical trial drug compared to baseline

SECONDARY OUTCOMES:
Change in Spherical Equivalent | 4, 8 months
  Change in spherical equivalent measured by cycloplegic autorefraction at 4, 8 months after administration of clinical trial drug compared to baseline
Change in Axial length (mm) | 4, 8, 12 months
  Change in Axial length (mm) at 4, 8, 12 months after administration of clinical trial drug compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Sei Yeul Oh, Principal Investigator — Samsung Medical Center
Locations (15):
- South Korea (15):
  - Pusan National University Hospital, Busan
  - Inje University Busan Paik Hospital, Busan
  - Kangwon National University Hospital, Chuncheon
  - Chungnam National University Hospital, Daejeon
  - Chung-Ang University Gwang Myeong hospital, Gwangmyeong
  - Gachon University Gil Hospital, Incheon
  - HanGil Eye Hospital, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si
  - Kim'S Eye Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul Asan Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul
  - Ajou University Hospital, Suwon
  - Yongin Severance Hospital, Yŏngin

IPD SHARING:
Plan to Share IPD: No